CLINICAL TRIAL: NCT03223818
Title: The Impact of Fast-track Perioperative Program on the Clinical and Immunological Outcomes After Liver Resection in Hong Kong Chinese Patients: A Prospective Randomized Trial
Brief Title: The Impact of Fast-track Perioperative Program After Liver Resection in Hong Kong Chinese Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Charing Chong, MD, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Fast-track_Liver Resection
Record Dates: First submitted 2015-11-11; First posted 2017-07-21 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Liver Cancer
Keywords: Liver; Digestive system
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fast-track Arm (Experimental): Patients recruited will undergo ERAS perioperative program.
  Interventions: Other: Fast-track peri-operative program
- Conventional Group (No Intervention): Patients recruited to conventional group will undergo conventional perioperative program

INTERVENTIONS:
Other: Fast-track peri-operative program — Patients who are scheduled for elective liver resection will be screened in clinic or in wards for the eligibility for ERAS program. Patient will then visit a nurse-led clinic for pre-operative assessment of risk adjustment and education. A guided tour on surgical ward and an information booklet about preoperative management will be given.
  All patients will receive local infiltration of local anaesthesia (0.25% levobupivacaine) followed by continuous wound instillation using the On-Q PainBuster System balloon pump. Pain control will be supplemented by using opioid-sparing multimodal analgesia.
  Other Names: Enhanced recovery after surgery(ERAS) peri-operative program
  Arms: Fast-track Arm

SUMMARY:
Liver cancer was the third leading cause of cancer death in both sexes in Hong Kong and liver resection remains the mainstay of curative treatment. Post-operative recovery from liver resection has historically been fraught with a high incidence of complications, ranging from 15-48%, and the high incidence of complications leads to prolonged hospital stay, ranging from 9 - 15 days, and increase costs of hospitalization. Recent advancement in the perioperative surgical and anesthetic management of patients undergoing liver resection has led to improvement in these outcomes.

The investigators department had previously studied the impact and confirmed the benefit of fast-track peri-operative programs after laparoscopic colorectal surgery. Nevertheless, studies regarding its adoption in liver resection are limited. The investigators group had previously reported, in a retrospective cohort, that successful implementation of ERAS protocol was associated with a significantly shorten hospital stay. However, the peri-operative management in that study incorporated a small proportion of components described in ERAS programs for liver resection and there was no direct comparison with conventional peri-operative program.

The aim of this study is to compare the clinical and immunological outcomes of Hong Kong Chinese patients undergoing liver resection for liver cancer with a "conventional" vs a "fast-track" perioperative program.

DETAILED DESCRIPTION:
Liver cancer was the third leading cause of cancer death in both sexes in Hong Kong and liver resection remains the mainstay of curative treatment. Post-operative recovery from liver resection has historically been fraught with a high incidence of complications, ranging from 15-48%, and the high incidence of complications leads to prolonged hospital stay, ranging from 9 - 15 days, and increase costs of hospitalization. Recent advancement in the perioperative surgical and anesthetic management of patients undergoing liver resection has led to improvement in these outcomes.

Since its formal introduction in 1990s, fast-track or enhanced recovery after surgery (ERAS) peri-operative programs have gained territory quickly because of the associated cost efficiency derived from the reduction in hospital stay, an important issue in today's context of rapidly increasing health care costs and the consequent need for optimization. The benefits of fast-track peri-operative programs have been well proven in colectomy. Our department had previously demonstrated the feasibility and impact of fast-track peri-operative programs after laparoscopic colorectal surgery, which leads to the potential for application to other subspecialties. Nevertheless, studies evaluating fast-track peri-operative programs in liver resection are scarce. Most of them were carried out in Western countries and almost all of them used epidural analgesia for post-operative pain control. While most of the livers in Western patients are non-cirrhotic, the main challenge of liver resection in Chinese Hong Kong patients is the background liver cirrhosis as hepatitis-related hepatocellular carcinoma is the most common indication for liver resection. Although epidural analgesia has been showed to be effective after liver resection without complication, the debate on epidural analgesia continues. Coagulopathy, thrombocytopenia and other haematological abnormalities may impose additional risks of epidural hematoma formation following removal of the epidural catheter postoperatively. Especially there is a much greater incidence of co-existing liver cirrhosis in Chinese Hong Kong patients with hepatocelluar carcinoma. This group of patients is coagulopathic even before liver resection and the risk of bleeding complications related to epidural analgesia is a particular concern. Continuous wound instillation with local anesthetic agent by the ON-Q PainBuster System (I-Flow Corporation, Lake Forest, CA, USA) provides an attractive alternative for this group of patients. We had previously demonstrated its analgesic efficacy after open hepatic surgery in a randomized controlled trial. Recently, our group had reported, in a retrospective cohort, that successful implementation of ERAS protocol was associated with a significantly shorten hospital stay. However, there was no direct comparison with convention peri-operative program in a randomized controlled manner. Moreover, the peri-operative management in that study incorporated only a small proportion of components described in ERAS programs for liver surgery, namely pre-operative counselling, no premedication, normothermia during surgery, no nasogastric tube and no routine abdominal drain. Furthermore, patient-controlled morphine analgesia was the method for post-operative pain control, which might not be enough for open hepatectomy and might have restricted the mobilization.

ELIGIBILITY:
Inclusion Criteria:

1. All consecutive patients undergoing elective liver resection (open and laparoscopic).
2. Age of patients between 18 and 70 years.
3. Patients with American Society of Anaesthesiologists (ASA) grading I-II.
4. Patients with no severe physical disability.
5. Patients who require no assistance on the activities of daily living.
6. Informed consent available will be recruited.

Exclusion Criteria:

1. Patients undergoing emergency surgery.
2. Patients who had received pre-operative portal vein embolization.
3. Patients who are expected to receive concomitant procedures other than cholecystectomy.
4. Pregnant ladies and patients who are mentally incapable of written consent will be excluded.
5. Patient who had previous history of Hepato-biliary and pancreatic surgery.
6. Patient who had chronic pain syndrome.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Length of post-operative hospital Stay | 3 months
  Post-operative hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No